CLINICAL TRIAL: NCT04746482
Title: Outcome of Root Canal Retreatment Performed in Single Visits. A Retrospective Study
Brief Title: Retrospective Assessment of Root Canal Retreatment Performed in Single Visit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dubai Health Authority (Other Government)
Responsible Party: Principal Investigator, Hend Mahmoud Abou El Nasr, Associate Professor/Specialist Senior Registrar, Dubai Health Authority
Other Study IDs: DSREC-01/2021_11
Record Dates: First submitted 2021-01-31; First posted 2021-02-09 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Root Canal Retreatment
Keywords: retrospective study; single visit; root canal retreatment; outcome; clinical; radiographic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- exposure group: subjects in this group are single visit
  Interventions: Procedure: single visit root canal retreatment

INTERVENTIONS:
Procedure: single visit root canal retreatment — cases that were subject to root canal retreatment performed in single visit

SUMMARY:
In cases refractory to initial root canal therapy in which a decision is made to perform nonsurgical retreatment, the patient has the right to know the prognosis of the proposed treatment and clinicians must be able to provide this information based on the best available data. The literature answered this question when the treatment was performed in multiple visits; however, little information exists when single visit root canal retreatment was performed. Therefore, the aim of the present study is to assess the clinical and radiographic outcome of root canal retreatment performed in single visits in endodontic clinics of Dubai Health Authority (DHA).

DETAILED DESCRIPTION:
The present study is designed to assess the clinical and radiographic outcome of root canal retreatment performed in single visits in endodontic clinics of Dubai Health Authority (DHA). This is a retrospective study where patients' treatment data will be collected and outcome criteria will be applied blindly.

The sample in this retrospective study will be selected from those patients who have undergone single visit endodontic retreatment at the DHA Endodontics clinics from January 2018, through December 2019. The teeth under investigation will be tracked in the database starting from completion of retreatment for at least 6 months, and the percentages of teeth that were retained or underwent additional procedures such as apical surgery or extraction will be recorded.

The clinical and radiographic assessment at baseline and at recall documented in clinical notes, and all data will be collected using a standardized proforma.

The quality of the existing root canal fillings and the status of the periapical tissues will be determined according to the PAI by 2 calibrated independent observers using the periapical radiographs.

A. Periapical index (PAI) The index is a radiographic method of interpretation that consists of 5 categories, numbered 1-5.

B. Quality of root canal filling

Three criteria were used to assess the quality of the existing root canal fillings as follows:

Length of root canal filling: root filling ending ≤2 mm from the radiographic apex, root filling ending >2 mm from the radiographic apex, or root filling at the radiographic apex (flush).

Density of root canal filling: the presence or absence of voids in the root filling or between the root filling and root canal walls.

Taper of the root canal filling: consistent taper from the orifice to the apex or no consistent taper from the orifice to the apex

The preoperative diagnosis is determined based on clinical and radiographic findings using the American Association of Endodontists Consensus Conference-recommended diagnostic terminology.

Retreatment Procedures

Endodontic retreatment of all cases was conducted in a single visit by endodontic specialists according to the contemporary standards of endodontic therapy.

Only those patients with at least 6 months of clinical and radiographic follow-up were included. When patients returned for recalls, one or multiple (in mutirooted teeth) periapical radiographs were taken.

Follow up

Recall appointments included a radiographic and clinical examination of the treated tooth. The examination was documented and included any signs or symptoms, the presence of a sinus tract, sensitivity to percussion and palpation, swelling, periodontal pockets, or a history of pain.

Periapical radiographs will be evaluated by 2 examiners.

The treatment outcomes will be classified into 3 categories according to the following definitions:

Healed: Functional, asymptomatic teeth with no or minimal radiographic periradicular pathosis (radiolucency) Nonhealed: Nonfunctional, symptomatic teeth with or without radiographic periradicular pathosis or asymptomatic teeth with unchanged, new, or enlarged radiographic periradicular pathosis (radiolucency) Healing: Teeth that are asymptomatic and functional with a decreased size of radiographic periradicular pathosis (radiolucency) .

Collecting data into a recording sheet:

The patients' treatment data will be collected continuously for at least 6 months in the database, and outcome criteria will applied blindly. The teeth will be tracked in the database during the entire period.

ELIGIBILITY:
Inclusion Criteria:

* Root canal retreatment cases performed in single visits
* Age ranging from 18 - 70 years
* Follow up period of at least 6 months

Exclusion Criteria:

A case will be excluded from the study if the case was under 18 years of age or followed up period for less than 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent root canal retreatment in single visit in endodontic clinics of Dubai Health Authority (DHA).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain or swelling | 6 months to 2 years
  dichotomized into yes or no
radiographic | 6 months to 2 years
  Periapical Index scoring scoring the health of the periapical area using a 5-scale scoring system (from 1 to 5); where1 represents normal periapical tissue while score 5 denotes established apical periodontitis

SECONDARY OUTCOMES:
Tooth survival | 6 months to 2 years
  Number of teeth retained or underwent additional procedures such as apical surgery and extraction

CONTACTS AND LOCATIONS:
Overall Officials: Hend Abou El Nasr, PhD, Principal Investigator — Cairo University and Dubai Health Authority
Locations (1):
- Dubai Health Authority, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Nuaimi N, Ciapryna S, Chia M, Patel S, Mannocci F. A prospective study on the effect of coronal tooth structure loss on the 4-year clinical survival of root canal retreated teeth and retrospective validation of the Dental Practicality Index. Int Endod J. 2020 Aug;53(8):1040-1049. doi: 10.1111/iej.13322. Epub 2020 Jun 8. PMID 32383194
- [Background] Habib AA, Doumani MD, Nassani MZ, Shamsy E, Jto BS, ArwadI HA, Mohamed SA. Radiographic Assessment of the Quality of Root Canal Fillings Performed by Senior Dental Students. Eur Endod J. 2018 Jul 19;3(2):101-106. doi: 10.14744/eej.2018.69775. eCollection 2018. PMID 32161864
- [Background] Eliyas S, Briggs PFA, Harris IR, Newton JT, Gallagher JE. Development of quality measurement instruments for root canal treatment. Int Endod J. 2017 Jul;50(7):652-666. doi: 10.1111/iej.12679. Epub 2016 Aug 19. PMID 27422536
- [Background] Goldberg F, Cantarini C, Alfie D, Macchi RL, Arias A. Relationship between unintentional canal overfilling and the long-term outcome of primary root canal treatments and nonsurgical retreatments: a retrospective radiographic assessment. Int Endod J. 2020 Jan;53(1):19-26. doi: 10.1111/iej.13209. Epub 2019 Sep 30. PMID 31454090
- [Background] Ng YL, Mann V, Gulabivala K. Outcome of secondary root canal treatment: a systematic review of the literature. Int Endod J. 2008 Dec;41(12):1026-46. doi: 10.1111/j.1365-2591.2008.01484.x. PMID 19133093
- [Background] Gorni FG, Gagliani MM. The outcome of endodontic retreatment: a 2-yr follow-up. J Endod. 2004 Jan;30(1):1-4. doi: 10.1097/00004770-200401000-00001. PMID 14760899
- [Background] de Chevigny C, Dao TT, Basrani BR, Marquis V, Farzaneh M, Abitbol S, Friedman S. Treatment outcome in endodontics: the Toronto study--phases 3 and 4: orthograde retreatment. J Endod. 2008 Feb;34(2):131-7. doi: 10.1016/j.joen.2007.11.003. Epub 2007 Dec 21. PMID 18215667
- [Background] Erdem Hepsenoglu Y, Eyuboglu TF, Ozcan M. Postoperative Pain Intensity after Single- versus Two-visit Nonsurgical Endodontic Retreatment: A Randomized Clinical Trial. J Endod. 2018 Sep;44(9):1339-1346. doi: 10.1016/j.joen.2018.05.017. Epub 2018 Jul 24. PMID 30054099
- [Background] Eyuboglu TF, Olcay K, Ozcan M. A clinical study on single-visit root canal retreatments on consecutive 173 patients: frequency of periapical complications and clinical success rate. Clin Oral Investig. 2017 Jun;21(5):1761-1768. doi: 10.1007/s00784-016-1957-2. Epub 2016 Sep 22. PMID 27660159
- [Background] Yoldas O, Topuz A, Isci AS, Oztunc H. Postoperative pain after endodontic retreatment: single- versus two-visit treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Oct;98(4):483-7. doi: 10.1016/j.tripleo.2004.03.009. PMID 15472665